CLINICAL TRIAL: NCT00485316
Title: Prospective Randomized Trial Comparing Laparoscopic Assisted and Open Resection for Colonic and Rectal Carcinoma
Brief Title: Laparoscopic Assisted Versus Open Resection for Colorectal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Ka Lau Leung, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-8118
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Colorectal Carcinoma
Keywords: Colorectal carcinoma; Rectal carcinoma; Laparoscopy; Laparoscopic surgery; Open surgery; Randomized trial
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Laparoscopic assisted resection of colorectal carcinoma

SUMMARY:
The aim of the investigators' randomized trial is to compare the short-term clinical outcome and survival between laparoscopic-assisted and open resection of colorectal carcinoma.

DETAILED DESCRIPTION:
Since the introduction of laparoscopic cholecystectomy in 1987, laparoscopic surgery has been attempted and applied to many surgical operations. Surgeons in Hong Kong began to perform laparoscopic surgery for colorectal carcinoma in early 1992. Early reports of laparoscopic surgery for colorectal carcinoma from Hong Kong and worldwide suggested better short-term clinical outcomes when compared with open surgery, but there were concerns over port site metastases and adequacy of long-term oncological clearance. Besides, only a few randomized trials thus far have compared laparoscopic-assisted and open surgery for rectal carcinoma.

The aim of our randomized trial is to compare the short-term clinical outcome and survival between laparoscopic-assisted and open resection of colonic and rectal carcinoma.

Patients will undergo different types of surgery according to the location of the tumors: right or extended right hemicolectomy for cecal, ascending colon, or hepatic flexure tumors; left hemicolectomy for descending colon tumors; sigmoid colectomy for sigmoid colon tumors; anterior resection for rectosigmoid or upper rectal tumors; low anterior resection with total mesorectal excision for mid- and low rectal tumors; abdominoperineal resection for very low rectal tumors. Patients will be randomly allocated to laparoscopic assisted or conventional open surgery.

Short-term clinical outcome and long-term survival data will be prospectively recorded and compared between the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed to have colorectal carcinoma at all locations except transverse colon
* Informed consent available

Exclusion Criteria:

* Patients with tumor >6 cm in size, or with tumor infiltration to adjacent organs on imagings
* Patients with previous abdominal surgery near the region of the colorectal surgery
* Patients with intestinal obstruction or perforation
* Patients with recurrent disease
* Patients with synchronous colorectal carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Overall survival and disease-free survival

SECONDARY OUTCOMES:
Operative time
Blood loss
Postoperative analgesic requirements
Recovery of gastrointestinal function (time to resume normal diet, time first passing flatus, time of first bowel motion)
Time to walk independently
Duration of hospital stay
Morbidity and mortality
Direct cost

CONTACTS AND LOCATIONS:
Overall Officials: Ka Lau Leung, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong SAR, China

REFERENCES:
- [Derived] Ng SS, Lee JF, Yiu RY, Li JC, Hon SS, Mak TW, Ngo DK, Leung WW, Leung KL. Laparoscopic-assisted versus open total mesorectal excision with anal sphincter preservation for mid and low rectal cancer: a prospective, randomized trial. Surg Endosc. 2014 Jan;28(1):297-306. doi: 10.1007/s00464-013-3187-x. Epub 2013 Sep 7. PMID 24013470
- [Derived] Li JC, Leung KL, Ng SS, Liu SY, Lee JF, Hon SS. Laparoscopic-assisted versus open resection of right-sided colonic cancer--a prospective randomized controlled trial. Int J Colorectal Dis. 2012 Jan;27(1):95-102. doi: 10.1007/s00384-011-1294-5. Epub 2011 Aug 23. PMID 21861071